CLINICAL TRIAL: NCT01275924
Title: Tightrope or Screw Fixation of Acute Tibiofibular Syndesmotic Injury. Randomised Controlled Trial.
Brief Title: Tightrope or Screw Fixation of Acute Tibiofibular Syndesmotic Injury
Acronym: TIGHTROPE-SS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset Asker og Baerum (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Wender Figved, MD PhD, Sykehuset Asker og Baerum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TIGHTROPE-SS
Record Dates: First submitted 2011-01-11; First posted 2011-01-13 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Syndesmotic Injury of the Ankle
Keywords: Syndesmosis; Injury; Ankle; Fracture
MeSH Terms: conditions — Wounds and Injuries; Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tightrope (Active Comparator): Treatment with Tightrope Syndesmosis Repair Kit
  Interventions: Device: Tightrope Syndesmosis Repair Kit
- Syndesmotic screw (Active Comparator): Treatment with a quadricortical syndesmotic screw
  Interventions: Device: Syndesmotic screw

INTERVENTIONS:
Device: Tightrope Syndesmosis Repair Kit — Tightrope Syndesmosis Repair Kit
  Other Names: Tightrope Syndesmosis Repair Kit, Arthrex; Naples, Florida
  Arms: Tightrope
Device: Syndesmotic screw — Quadricortical syndesmotic screw
  Other Names: Cortical screw; Synthes GmbH, Switzerland
  Arms: Syndesmotic screw

SUMMARY:
Syndesmotic injuries are common and often associated with unstable ankle fractures. The most common treatment is with a syndesmotic screw through the fibula and tibia which is later removed, usually after 10-12 weeks. The Tightrope Syndesmosis Repair Kit (Arthrex; Naples, Florida). is used for the same indication, it consists of a heavy suture placed across the syndesmosis which has been looped and tightened through cortical button anchors on either side of the ankle. It does not need removal and thus avoids subsequent surgery. This trial compares these two treatment methods for syndesmotic injuries of the ankle.

DETAILED DESCRIPTION:
Patients 18-70 years presenting to one of the two hospitals with an acute syndesmotic injury are eligible for inclusion. 50 patients are randomised to two treatment groups: One group receives a Tightrope (R) fixation and the other receives a quadricortical screw fixation which is removed after 12 weeks. Follow-up intervals are at 6 weeks, 6, 12 and 24 months with standardised CT scans postoperatively and at 12, 24 months and 5 years clinical end-ponts/scores.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years
* Acute syndesmotic injury with or without Weber type C fracture

Exclusion Criteria:

* Prior injury of the same ankle
* Severe injury of same leg affecting rehabilitation
* Symptomatic osteoarthritis of same ankle
* Open injury
* Decubital injury affecting surgical site
* Dementia or unable to sign informed consent
* Neuropathic conditions affecting same leg

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2011-01; Primary Completion 2015-03 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
OTA Score (Modified American Orthopaedic Foot and Ankle Society ankle hind foot score) | 5 years
  Modified American Orthopaedic Foot and Ankle Society ankle hind foot score (0-100)

SECONDARY OUTCOMES:
Olerud-Molander Ankle (OMA) Score | 5 years
Dorsiflexion angle | 5 years
  According to Lindsjø
Health-related quality of life (EQ-5D) | 5 years
CT measurements of syndesmotic distance | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Wender Figved, MD, PhD, Study Director — Baerum Hospital, Vestre Viken, Norway
Locations (2):
- Norway (2):
  - Oslo University Hospital, Oslo
  - Baerum Hospital, Vestre Viken, Rud